CLINICAL TRIAL: NCT07250802
Title: A Phase 3, Randomized, Multicenter, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Zasocitinib in Pediatric Participants Aged 4 to Less Than 18 Years With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Long-Term Study of Zasocitinib in Children and Teenagers With Plaque Psoriasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-279-PsO-3006; 2025-522567-15-00 (EU CTIS Number); jRCT2071250114 (Registry Identifier: jRCT)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part A: Double-blinded and Open-label; Part B: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A (Cohort 1): Zasocitinib (Dose A) (Experimental): Participants (Adolescent) aged 12 to less than (<)18 years will receive zasocitinib Dose A once daily (QD), orally, from Week 1 to Week 16 during the double-blind placebo-controlled period followed by zasocitinib, from Week 16 to Week 208 during the open-label period.
  Interventions: Drug: Zasocitinib
- Part A (Cohort 2): Zasocitinib (Multiple Doses) (Experimental): Participants (Children) aged 4 to <12 years will receive zasocitinib, orally, doses based on weight, from Week 1 to Week 16 during the double-blind placebo-controlled period followed by zasocitinib from Week 16 to Week 208 during the open-label period.
  Interventions: Drug: Zasocitinib
- Part A (Cohort 1 and Cohort 2): Placebo (Placebo Comparator): Participants in Cohort 1 (Adolescent aged 12 to <18 years) and Cohort 2 (Children aged 4 to <12 years) will receive zasocitinib matching placebo QD from Week 1 to Week 16 during the double-blind placebo-controlled period.
  Interventions: Drug: Placebo
- Part B: Zasocitinib (Multiple Doses) (Experimental): Participants (Children) aged 4 to <12 years will receive zasocitinib, orally, doses based on weight, from Week 1 to Week 208 during the open-label period.
  Interventions: Drug: Zasocitinib

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib.
  Other Names: TAK-279; NDI-034858
  Arms: Part A (Cohort 1): Zasocitinib (Dose A)
Drug: Placebo — Zasocitinib matching placebo.
  Arms: Part A (Cohort 1 and Cohort 2): Placebo
Drug: Zasocitinib — Zasocitinib.
  Other Names: TAK-279; NDI-034858
  Arms: Part A (Cohort 2): Zasocitinib (Multiple Doses); Part B: Zasocitinib (Multiple Doses)

SUMMARY:
The main aim of this study is to see how well the medicine zasocitinib works, how safe it is, and how children and teenagers aged 4 to under 18 with moderate-to-severe plaque psoriasis respond to it.

The study will be done in 2 parts: Part A will include both children and teenagers, while part B will only include children.

At first, only teenagers who meet the study rules can participate in this study. Children may only start to participate once enough information has been collected from other studies with zasocitinib.

Participants in Part A will initially be assigned to receive either zasocitinib or placebo for the first 16 weeks of treatment, then all participants will receive zasocitinib through the end of the study. All participants in Part B will be assigned to receive treatment with zasocitinib throughout the study.

Participants will be in the study for up to 4 years and 2 months (217 weeks), including up to 35 days for the screening period, 208 weeks of treatment (Part A and Part B) and a 4-week safety follow-up period. During the study, participants will visit their study site multiple times.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a diagnosis of chronic plaque psoriasis for greater than or equal to (>=) 6 months prior to the screening visit.
2. Participant has stable plaque psoriasis defined as no significant flare or change in morphology (as assessed by the investigator) in psoriasis for >=6 months before screening.
3. Participant has moderate-to-severe plaque psoriasis as defined by a Psoriasis Area and Severity Index (PASI) score >=12 and a Static Physician's Global Assessment (sPGA) score >=3 at screening and Day 1.
4. Participant has plaque psoriasis covering >=10 percent (%) of total body surface area (BSA) at screening and Day 1.
5. Participant must be a candidate for phototherapy or systemic therapy.
6. Inclusion Criteria for Part A Cohort 1: The participant is male or female and aged 12 to less than (<) 18 years, inclusive.
7. Inclusion Criteria for Part A Cohort 2 and for Part B: The participant is male or female and aged 4 to <12 years, inclusive.
8. Inclusion Criteria for Part A Cohort 1: The participant must weigh >=40 kilograms (kg) at the time of screening.

Exclusion Criteria:

1. Participant has evidence of nonplaque psoriasis (erythrodermic, pustular, predominantly guttate psoriasis, predominantly inverse, or drug-induced psoriasis). If a participant meets criteria for inclusion based on typical plaque psoriasis presentation, a limited amount of inverse psoriasis is not exclusionary.
2. Participant requires systemic treatment, other than nonsteroidal anti-inflammatory drugs (NSAIDs), during the trial period for an immune-related disease.
3. Participant has concomitant comorbid skin condition that, in the opinion of the investigator, would interfere with the trial assessments.
4. Participant has history of active TB infection, regardless of treatment status and has signs or symptoms of active TB or evidence of latent tuberculosis infection (LTBI).
5. Participant has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 or a history of serious herpetic infection.
6. Participant has a history of chronic or recurrent bacterial disease.
7. Participant has a history of opportunistic infections (for example, Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
8. Participant has any clinically significant medical condition, evidence of an unstable clinical condition or vital signs/physical examination/laboratory/ECG abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of trial results.
9. Participant has any previous exposure to zasocitinib (also known as TAK-279 or NDI-034858) or other TYK2 inhibitors or participated in any trial that included a tyrosine kinase 2 (TYK2) inhibitor, unless participant has documentation of posttrial unblinding that confirms the participant did not receive a TYK2 inhibitor.
10. Participant is not up to date on all required vaccinations according to current immunization guidelines as noted by country-specific pediatric authorities.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2033-01-24 (Estimated); Study Completion 2033-01-24 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants Achieving a Static Physician's Global Assessment (sPGA) of Clear (0) or Almost Clear (1) With a Greater than or Equal to (>=) 2-Point Decrease From Baseline at Week 16 | At Week 16
  The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean greater than (>) 0, less than (<) 1.5; Mild (2) = mean >= 1.5, <2.5; Moderate (3) = mean >=2.5, <3.5; and Severe (4) = mean >=3.5. The percentage of participants achieving an sPGA of Clear (0) or Almost Clear (1) with a >= 2-point decrease from baseline at Week 16 will be reported.
Part A: Percentage of Participants Achieving >= 75 Percent (%) Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 16 | At Week 16
  The PASI is a measure of the average redness, thickness and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity (less than or equal to [<=] 3 representing mild disease, >= 3 to 15 representing moderate disease, and >= 15 indicating severe disease). The PASI-75 is defined as 75% improvement from baseline in PASI score. The percentage of participants achieving >= 75% improvement from baseline in PASI score at Week 16 will be reported.
Part B: Maximum Observed Plasma Concentration (Cmax) of Zasocitinib | Pre-dose and Post-dose on Day 7
  Cmax of zasocitinib in plasma will be assessed.
Part B: Time to Maximum Concentration (Tmax) of Zasocitinib | Pre-dose and Post-dose on Day 7
  Tmax of zasocitinib in plasma will be assessed.
Part B: Area Under the Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-Last) of Zasocitinib | Pre-dose and Post-dose on Day 7
  AUC0-Last of zasocitinib in plasma will be assessed.

SECONDARY OUTCOMES:
Part A: Percentage of Participants Achieving PASI-90 Response at Week 16 | At Week 16
  The PASI is a measure of the average redness, thickness and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity (less than or equal to [<=] 3 representing mild disease, >= 3 to 15 representing moderate disease, and >= 15 indicating severe disease). The PASI-90 is defined as 90% improvement from baseline in PASI score. The percentage of participants achieving at least 90% or greater reduction in the PASI score from baseline at Week 16 will be assessed.
Part A: Percentage of Participants Achieving an Enhanced sPGA Response of Clear (0) at Week 16 | At Week 16
  The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean greater than (>) 0, less than (<) 1.5; Mild (2) = mean >= 1.5, <2.5; Moderate (3) = mean >=2.5, <3.5; and Severe (4) = mean >=3.5. The percentage of participants achieving an enhanced sPGA response of Clear (0) at Week 16 will be assessed.
Part A: Percentage of Participants Achieving PASI-100 Response at Week 16 | At Week 16
  The PASI is a measure of the average redness, thickness and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity (less than or equal to [<=] 3 representing mild disease, >= 3 to 15 representing moderate disease, and >= 15 indicating severe disease). The PASI-100 is defined as 100% improvement from baseline in PASI score. The percentage of participants achieving 100% improvement or complete clearance of psoriasis lesions in the PASI score from baseline at Week 16 will be assessed.
Part A: Percentage of Participants Achieving a Scalp-specific Physician's Global Assessment (ssPGA) Response of Clear (0) or Almost Clear (1) With a >=2-Point Decrease From Baseline for Participants With a Baseline ssPGA >=3 at Week 16 | At Week 16
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate more severe scalp psoriasis. The percentage of participants achieving an ssPGA score of at least 3 at baseline who show an ssPGA score of 0 or 1 with a >= 2-point decrease at Week 16 will be reported.
Part A: Change From Baseline in Body Surface Area (BSA) Affected by Psoriasis at Week 16 | Baseline, Week 16
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement. The change from baseline in BSA affected by psoriasis at Week 16 will be assessed.
Part A: Percent Change From Baseline in BSA Affected by Psoriasis at Week 16 | Baseline, Week 16
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement. The percent change from baseline in BSA affected by psoriasis at Week 16 will be assessed.
Part A: Percentage of Participants with a Baseline Dermatology Life Quality Index (DLQI) Score >=2 who Achieve DLQI Score of Zero (0) or One (1) at Week 16 | At Week 16
  The DLQI is a 10-item validated questionnaire completed by participants aged 16 years or older at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life). The percentage of participants with a baseline DLQI Score >= 2 who achieve DLQI Score of Zero (0) or One (1) at Week 16 will be assessed.
Part A: Percentage of Participants With a Baseline Children's Dermatology Life Quality Index (CDLQI) Score >=2 who Achieve CDLQI Score of 0 or 1 at Week 16 | At Week 16
  The CDLQI is a 10-item validated questionnaire completed by participants aged 4 to <16 years of age at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains designed to measure the impact of skin disease on the child's quality of life, including symptoms and feelings, daily activities, leisure, school, personal relationships and treatment. The CDLQI score ranges from 0 to 30 points, higher score indicates greater severity. The percentage of participants with a baseline CDLQI Score >=2 who achieve CDLQI Score of 0 or 1 at Week 16 will be assessed.
Part A: Change From Baseline in DLQI at Week 16 | Baseline, Week 16
  The DLQI is a 10-item validated questionnaire completed by participants aged 16 years or older at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life). The change from baseline in DLQI at Week 16 will be assessed.
Part A: Change From Baseline in CDLQI at Week 16 | Baseline, Week 16
  The CDLQI is a 10-item validated questionnaire completed by participants aged 4 to <16 years of age at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains designed to measure the impact of skin disease on the child's quality of life, including symptoms and feelings, daily activities, leisure, school, personal relationships and treatment. The CDLQI score ranges from 0 to 30 points, higher score indicates greater severity. The change from baseline in CDLQI at Week 16 will be assessed.
Part A (Cohort 1): Percentage of Participants in Cohort 1 with a Baseline Itch Numerical Rating Scale (NRS) Score >=4 who Achieve a >= 4-Point Improvement in Itch NRS Score at Week 16 | At Week 16
  The Itch NRS is a single-item participant-reported measure. Participants indicate itch severity at its worst over a 24-hour recall period on an 11-point scale anchored at 0, representing 'no itching' and 10, representing 'worst itch imaginable'. The percentage of participants in Cohort 1 with a baseline Itch NRS Score >=4 who achieve a >=4-Point improvement in Itch NRS Score at Week 16 will be assessed.
Part A (Cohort 1): Change From Baseline in Itch NRS at Week 16 | Baseline, Week 16
  The Itch NRS is a single-item participant-reported measure. Participants indicate itch severity at its worst over a 24-hour recall period on an 11-point scale anchored at 0, representing 'no itching' and 10, representing 'worst itch imaginable'. The change from baseline in Itch NRS at Week 16 will be assessed.
Part A (Cohort 1): Percent Change From Baseline in Itch NRS at Week 16 | Baseline, Week 16
  The Itch NRS is a single-item participant-reported measure. Participants indicate itch severity at its worst over a 24-hour recall period on an 11-point scale anchored at 0, representing 'no itching' and 10, representing 'worst itch imaginable'. The percent change from baseline in Itch NRS at Week 16 will be assessed.
Parts A and B: Percentage of Participants Achieving PASI-75 Response During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The PASI is a measure of the average redness, thickness and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity (less than or equal to [<=] 3 representing mild disease, >= 3 to 15 representing moderate disease, and >= 15 indicating severe disease). The PASI-75 is defined as 75% improvement from baseline in PASI score. The percentage of participants achieving at least 75% or greater reduction in the PASI score from baseline during open-label period will be reported.
Parts A and B: Percentage of Participants Achieving PASI-90 During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The PASI is a measure of the average redness, thickness and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity (less than or equal to [<=] 3 representing mild disease, >= 3 to 15 representing moderate disease, and >= 15 indicating severe disease). The PASI-90 is defined as 90% improvement from baseline in PASI score. The percentage of participants achieving at least 90% or greater reduction in the PASI score from baseline during open-label period will be reported.
Parts A and B: Percentage of Participants Achieving PASI-100 During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The PASI is a measure of the average redness, thickness and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI score ranges from 0 to 72, with higher PASI scores denoting more severe disease activity (less than or equal to [<=] 3 representing mild disease, >= 3 to 15 representing moderate disease, and >= 15 indicating severe disease). The PASI-100 is defined as 100% improvement from baseline in PASI score. The percentage of participants achieving 100% improvement or complete clearance of psoriasis lesions in the PASI score from baseline during open-label period will be reported.
Parts A and B: Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) With a >=2-Point Decrease From Baseline | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean greater than (>) 0, less than (<) 1.5; Mild (2) = mean >= 1.5, <2.5; Moderate (3) = mean >=2.5, <3.5; and Severe (4) = mean >=3.5. The percentage of participants achieving an sPGA of Clear (0) or Almost Clear (1) with a >=2-point decrease from baseline will be reported.
Parts A and B: Percentage of Participants Achieving an Enhanced sPGA of Clear (0) During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean greater than (>) 0, less than (<) 1.5; Mild (2) = mean >= 1.5, <2.5; Moderate (3) = mean >=2.5, <3.5; and Severe (4) = mean >=3.5. The percentage of participants achieving an enhanced sPGA of Clear (0) during open-label period will be reported.
Parts A and B: Percentage of Participants Achieving an ssPGA Response of Clear (0) or Almost Clear (1) with a >=2-point Decrease From Baseline for Participants with a Baseline ssPGA >=3 During Open-Label Period | Part A: Week 16 to Week 208
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate more severe scalp psoriasis. The percentage of participants achieving an ssPGA response of clear (0) or almost clear (1) with a >=2-point decrease from baseline for participants with a baseline ssPGA >=3 during open-label period will be reported.
Parts A and B: Change From Baseline in BSA Affected by Psoriasis During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement. The change from baseline in BSA affected by psoriasis during open-label period will be assessed.
Parts A and B: Percent Change From Baseline in BSA Affected by Psoriasis During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement. The percent change from baseline in BSA affected by psoriasis during open-label period will be assessed.
Parts A and B: Percentage of Participants With a Baseline DLQI Score >=2 who Achieve DLQI Score of 0 or 1 During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The DLQI is a 10-item validated questionnaire completed by participants aged 16 years or older at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life). The percentage of participants with a baseline DLQI Score >= 2 who achieve DLQI Score of 0 or 1 during open-label period will be assessed.
Parts A and B: Percentage of Participants With a Baseline CDLQI Score >=2 who Achieve CDLQI Score of 0 or 1 During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The CDLQI is a 10-item validated questionnaire completed by participants aged 4 to <16 years of age at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains designed to measure the impact of skin disease on the child's quality of life, including symptoms and feelings, daily activities, leisure, school, personal relationships and treatment. The CDLQI score ranges from 0 to 30 points, higher score indicates greater severity. The percentage of participants with a baseline CDLQI Score >= 2 who achieve CDLQI Score of 0 or 1 during open-label period will be assessed.
Parts A and B: Change From Baseline in DLQI During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The DLQI is a 10-item validated questionnaire completed by participants aged 16 years or older at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life). The change from baseline in DLQI during open-label period will be assessed.
Parts A and B: Change From Baseline in CDLQI During Open-Label Period | Part A: Week 16 to Week 208; Part B: Week 1 to Week 208
  The CDLQI is a 10-item validated questionnaire completed by participants aged 4 to <16 years of age at screening, which is used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The questionnaire covers 6 domains designed to measure the impact of skin disease on the child's quality of life, including symptoms and feelings, daily activities, leisure, school, personal relationships and treatment. The CDLQI score ranges from 0 to 30 points, higher score indicates greater severity. The change from baseline in CDLQI during open-label period will be assessed.
Part A (Cohort 1): Percentage of Participants with a Baseline Itch Numerical Rating Scale (NRS) Score >=4 who Achieve a >= 4-Point Improvement in Itch NRS Score During Open-Label Period | Part A: Week 16 to Week 208
  The Itch NRS is a single-item participant-reported measure. Participants indicate itch severity at its worst over a 24-hour recall period on an 11-point scale anchored at 0, representing 'no itching' and 10, representing 'worst itch imaginable'. The percentage of participants with a baseline Itch NRS score >=4 who achieve a >=4-Point improvement in Itch NRS score during open-label period will be assessed.
Part A (Cohort 1): Change From Baseline in Itch NRS for Participants in Cohort 1 During Open-Label Period | Part A: Baseline, Week 16 to Week 208
  The Itch NRS is a single-item participant-reported measure. Participants indicate itch severity at its worst over a 24-hour recall period on an 11-point scale anchored at 0, representing 'no itching' and 10, representing 'worst itch imaginable'. The change from baseline in Itch NRS for participants in Cohort 1 during open-label period will be assessed.
Part A (Cohort 1): Percent Change From Baseline in Itch NRS for Participants in Cohort 1 During Open-Label Period | Part A: Baseline, Week 16 to Week 208
  The Itch NRS is a single-item participant-reported measure. Participants indicate itch severity at its worst over a 24-hour recall period on an 11-point scale anchored at 0, representing 'no itching' and 10, representing 'worst itch imaginable'. The percent change from baseline in Itch NRS for participants in Cohort 1 during open-label period will be assessed.
Part A: Plasma Concentrations of Zasocitinib in Participants Receiving Active Treatment | Part A: Week 1 to Week 208
  Plasma concentrations of zasocitinib will be assessed using a validated liquid chromatography tandem mass spectrometry bioanalytical method.
Part B: Zasocitinib Acceptability and Palatability Assessment Scores of Participants | Day 1, Day 7 and Day 14
  The acceptability and palatability of zasocitinib will be assessed using the Acceptability Palatability Questionnaire. In this 5-item questionnaire, participants will be asked to evaluate the palatability and acceptability of zasocitinib considering the following elements: smell, taste, ease of swallowing, and aftertaste. This questionnaire uses an 11-point scale anchored at 0; a higher score means better acceptability and palatability.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (40):
- United States (11):
  - Exalt Clinical Research, Chula Vista, California
  - First OC Dermatology Research Inc., Fountain Valley, California
  - Direct Helpers Medical Center, Hialeah, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Apex Clinical Research Center, LLC, Canton, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Apex Clinical Research Center, LLC, Mayfield Heights, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Physicians Dermatology - Bellaire Station, Bellaire, Texas
  - Texas Dermatology and Laser Specialists-San Antonio, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- China (6):
  - Beijing Children Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hunan Children's Hospital, Changsha, Hunan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Peking University Third Hospital, Beijing
  - Huashan Hospital Fudan University, Shanghai
- Germany (6):
  - Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Uniklinik Koln, Klinik fur Dermatologie und Venerologie, Cologne, North Rhine-Westphalia
  - University Hospital of Muenster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn
  - Universitaetsmedizin der Johannes - Gutenberg Universitaet Mainz, Mainz
- Italy (3):
  - Presidio Ospedaliero Gaspare Rodolico, Catania, Sicily
  - Universita Degli Studi Di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Japan (5):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-shi, Fukuoka
  - Mie University Hospital, Tsu, Mie, Mie-ken
  - Nippon Life Hospital, Osaka, Osaka
  - Teikyo University Hospital, Itabashi-Ku, Tokyo
- Poland (6):
  - Cityclinic Przychodnia lekarsko psychologiczna Matusiak sp.p, Wroclaw, Lower Silesian Voivodeship
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Dorota Krasowska, Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Fryderyka Chopina w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - Centrum Badan Klinicznych Pi-house Sp. Z O. O., Gdansk, Pomeranian Voivodeship
  - "DERMED" Centrum Medyczne Sp. z o. o., Lodz
  - Dermoklinika-Centrum Medyczne s.c, Lodz
- Spain (3):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital de La Santa Creu i Sant Pau - Dermatologia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/2b154a9aa0bc4471??page=1&idFilter=TAK-279-PsO-3006